CLINICAL TRIAL: NCT03976453
Title: Psychological Outcome of Women With Morbidly Adherent Placenta Following Hystrectomy: Prospective Matched Case-control Study
Brief Title: Psychological Outcome of Women With Morbidly Adherent Placenta Following Hystrectomy
Status: Completed | Type: Observational
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Mostafa R Bakry, MBBCh, The principal investigator, Ain Shams Maternity Hospital
Other Study IDs: Morbidly Adherent Placenta
Record Dates: First submitted 2019-05-31; First posted 2019-06-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Morbidly Adherent Placenta
MeSH Terms: conditions — Placenta Accreta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: Women who underwent caesarean hysterectomy
- Group B: Women who underwent lower segment caesarean section
- Group C: Women who underwent spontaneous Vaginal delivery

SUMMARY:
The purpose of this study is to investigate the risk of postoperative psychiatric disorders of depression, anxiety outcomes and sexual dysfunctions and self esteem disturbance in women with morbidly adherent placenta following hysterectomy.

Research hypothesis:

In women with morbidly adherent placenta, We will predict, evaluate and decrease the psychological disorders following hysterectomy.

Research question:

Is there any difference in psychological outcome between caesarean section and caesarean hysterectomy ? This study aims to assess the psychological outcome in women with morbidly adherent placenta following hysterectomy.

DETAILED DESCRIPTION:
Morbidly adherent placenta, which describes placenta accreta, increta, and percreta, implies an abnormal implantation of the placenta into the uterine wall.

The incidence of placenta accreta has increased significantly over the past several decades, with the main risk factors include prior cesarean section and placental previa.

However, no well-designed trials have yet assessed the psychological outcome of women with morbidly adherent placenta following hystrectomy. The investigators will conduct a prospective matched case control trial to evaluate the psychological outcome to assess the risk of depression ,anxiety , sexual dysfunctions and self esteem disturbance following hysterectomy in women with morbidly adherent placenta.

This Prospective matched case-control trial will take place at Ain Shams University Maternity Hospital. Women in child bearing period, with morbidly adherent placenta will be eligible for inclusion.

Placenta accreta (Morbidly adherent placenta) is a condition in which all or part of the placenta is adherent to the uterine wall because of myometrial invasion by chorionic villi. It may occur when there is either a primary deficiency of or a secondary damage to chorionic villi or Nitabuch's layer.

Morbidly adherent placenta occurs in 5% of women with placenta previa. In some pregnancies, the placenta may develop at an abnormal location or may extensively invade the adjacent myometrium. Clinical entities include placenta previa, in which trophoblastic cells implant over or near the internal cervical os .In other cases, trophoblast aggressively burrows into the myometrium. Depending on the invasion depth, placenta accreta, placenta increta, or placenta percreta is diagnosed. The term placenta accrete syndromes is clinically useful to summarize these three types. Another interchangeable phrase also often used is morbidly adherent placenta .

Assisted reproductive technology and maternal smoking increase the risk of placenta.

The risk of accrete in women with a placenta previa and a prior caesarean section increased from 3% with one previous caesarean section to 11%, 40%, 61% and 67% with two, three, four, or more repeat caesarean sections respectively .

The maternal mortality risk may reach 7 % and the extensive surgery related morbidities include massive transfusions, infections, urologic injuries and fistula formation .

Women often consider the uterus to be a sexual organ, and the controller and regulator of important physiological functions in the body, as well as the source of youth, energy, activity, and a symbol of child-bearing capacity .

The relationship between hysterectomies and psychological disorders has been raised since the beginning of the 1990s. For example, in 1997, Thompson reported that there was a probability of psychoses in women after hysterectomies; and within the three years following the surgery, 33% of the women experienced symptoms of depression .

There are three broad subsets of psychological symptoms. These are: anxiety and depression attributed to the operation, sexual dysfunction (presenting as diminished libido, pain, dyspareunia or anxiety surrounding sexual activity) and reactions related to perceptions of feminity and low self-esteem.

ELIGIBILITY:
Inclusion Criteria:

- The 3 groups should be matched in age and parity. Age of child bearing period. Women who delivered from 4-6 months ago. At a gestational age after age of viability (28 weeks).

Exclusion Criteria:

- Pre-existing psychological disorders.

Max Age: 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Females in child bearing period
Study Population: Females in child bearing period presented with morbidly adherent placenta
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2019-06-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Depression | Baseline
  All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research through SCID I .Structured Clinical Interview for DSM-IV (SCID I) is a flexible semi structured diagnostic interview designed for use by trained clinicians to diagnose many adult DSM-IV axis I clinical disorders. It includes 7 diagnostic modules, focused on different diagnostic groups: mood, psychotic, substance abuse, anxiety, somatoform, eating and adjustment disorders then using Beck depression inventory scale.This is an inventory used for assessing the severity of depression state. It consists of 21 items, each of which has four responses of increasing severity. Numerical values from 0-3 are assigned each statement to indicate the degree of severity. The Arabic version will be used for the study.
Sexual dysfunction | Baseline
  All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research through a a test which is a brief questionnaire measure of sexual functioning in women. It is 19-item questionnaire has been developed as a multidimensional self-report instrument for assessing the key dimensions of sexual function in women. It provides scores on six domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction and pain) as well as a total score. The FSFI total score varies between 1.2 and 36, a score ≤ 26 defines sexual dysfunction. It is not a measure of sexual experience, knowledge, attitude, or interpersonal functioning in women. The Arabic version used in this research was a validated, reliable, and locally accepted tool for use in the assessment of female sexual disorder in the Egyptian population .
Anxiety | Baseline
  All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research through Taylor scale. It is performed to assess the anxiety state. This early instrument is derived from the MMPI in which the patient has to answer Yes or No to these questions, which are phrased in formal Arabic and can be understood by all those people who can read simple Arabic.
Self-esteem disturbance | Baseline
  All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research. The self esteem scale is an Arabic self reported questionnaire designed to assess the overall self esteem of the reporter. It measures the self view of the reporter to his capabilities in different situations, for example: social situations, interpersonal relations, future ambitions and previous accomplishments.
  It is composed of 30 items rated as follows: frequently = 2, sometimes = 1 and never = 0. Items indicating low self esteem are inversely scored. Scoring is done by summing the ordinary questions and inversely scored questions. Higher scores indicate higher self esteem.
  The instrument showed good internal consistency reliability (0.76). The construct convenient of the scale is fairly supported by factor analysis and convergent validation with other scales measuring self esteem

SECONDARY OUTCOMES:
Any other possible psychiatric morbidity | Baseline
  All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research through SCID I .Structured Clinical Interview for DSM-IV (SCID I) is a flexible semi structured diagnostic interview designed for use by trained clinicians to diagnose many adult DSM-IV axis I clinical disorders. It includes 7 diagnostic modules, focused on different diagnostic groups: mood, psychotic, substance abuse, anxiety, somatoform, eating and adjustment disorders. The Arabic version of the structured clinical interview for DSM-IV axis I (SCID-I) will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Amr El Shalakany, Prof, Principal Investigator — Ain Shams Maternity Hospital
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All data resulting from this study will be published
Supporting Information: Study Protocol
Time Frame: Baseline
Access Criteria: All patients will be subjected to fulfill Questionnaire after obtaining informed consent from the patients who are invited to participate in the research.

REFERENCES:
- [Background] Anis TH, Gheit SA, Saied HS, Al kherbash SA. Arabic translation of Female Sexual Function Index and validation in an Egyptian population. J Sex Med. 2011 Dec;8(12):3370-8. doi: 10.1111/j.1743-6109.2011.02471.x. Epub 2011 Oct 13. PMID 21995610
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Broome A and Wallace L, eds. (1984): Psychology and Gynecological Problems. Tavistock Publications, London.
- [Background] Cunningham FG, Leveno KJ, Bloom SL, et al. (eds) (2014): Obstetrical hemorrhage. In: Williams Obstetrics, 24th ed. New York, McGraw-Hill Education, pp: 505-511
- [Background] Cunningham FG, MacDonald PC, Gant NF et al. (eds) (1997): Obstetrical haemorrhage. In: Williams Obstetrics, 20th ed. Appleton& Lange: Stanford, CT, pp: 755-6.
- [Background] El Missiry A (2003): Homicide and psychiatric illness, An Egyptian study. MD Thesis, Faculty of Medicine, Ain Shams University.
- [Background] First MB, Spitzer RL and Williams W (1995): Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) in Handbook of Psychiatric Measures. Washington, American Psychiatric Association.
- [Background] Gielchinsky Y, Mankuta D, Rojansky N, Laufer N, Gielchinsky I, Ezra Y. Perinatal outcome of pregnancies complicated by placenta accreta. Obstet Gynecol. 2004 Sep;104(3):527-30. doi: 10.1097/01.AOG.0000136084.92846.95. PMID 15339763
- [Background] Jauniaux E, Alfirevic Z, Bhide AG, Belfort MA, Burton GJ, Collins SL, Dornan S, Jurkovic D, Kayem G, Kingdom J, Silver R, Sentilhes L; Royal College of Obstetricians and Gynaecologists. Placenta Praevia and Placenta Accreta: Diagnosis and Management: Green-top Guideline No. 27a. BJOG. 2019 Jan;126(1):e1-e48. doi: 10.1111/1471-0528.15306. Epub 2018 Sep 27. No abstract available. PMID 30260097
- [Background] O'Brien JM, Barton JR, Donaldson ES. The management of placenta percreta: conservative and operative strategies. Am J Obstet Gynecol. 1996 Dec;175(6):1632-8. doi: 10.1016/s0002-9378(96)70117-5. PMID 8987952
- [Background] Rahimzadeh A and Nazemi AR (2002): A Survey About the Effect Of Hysterectomy on Sexual Dysfunction in Patients Underwent Surgery in Sanandaj Behsat Hospital. Sci J Kurdistan Univ Med Sci; 2(3): 50-55.
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Silver RM, Landon MB, Rouse DJ, Leveno KJ, Spong CY, Thom EA, Moawad AH, Caritis SN, Harper M, Wapner RJ, Sorokin Y, Miodovnik M, Carpenter M, Peaceman AM, O'Sullivan MJ, Sibai B, Langer O, Thorp JM, Ramin SM, Mercer BM; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Maternal morbidity associated with multiple repeat cesarean deliveries. Obstet Gynecol. 2006 Jun;107(6):1226-32. doi: 10.1097/01.AOG.0000219750.79480.84. PMID 16738145
- [Background] TAYLOR JA. A personality scale of manifest anxiety. J Abnorm Psychol. 1953 Apr;48(2):285-90. doi: 10.1037/h0056264. No abstract available. PMID 13052352
- [Result] Alipour A and Pour Y (2010): Effect of cognitive behavioral therapy in hastening recovery of women after hysterectomy surgery. J Behav Sci; 4(2):91-5